CLINICAL TRIAL: NCT04058470
Title: Phase Ib/II Study of Toripalimab In Combination With Rituximab Followed by R-CHOP Regimen (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) for Elderly Naïve Patients With Diffuse Large B-cell Lymphoma
Brief Title: Toripalimab Plus Rituximab Followed by R-CHOP for Elderly Patients With Untreated Diffused B Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqiang Huang (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREND
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma Grade IIIb; Transformed Lymphoma; EBV-Positive DLBCL, Nos; ALK-Positive Anaplastic Large Cell Lymphoma
Keywords: DLBCL,HGL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic | interventions — toripalimab; Rituximab; R-CHOP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TR follow by R-CHOP (Experimental): TR follow by R-CHOP:
  TR: Toripalimab,Rituximab, R-CHOP: Rituximab, Cyclophosphamide,Doxorubicin,Vincristine,Prednisone
  Interventions: Drug: Toripalimab, Rituximab; Drug: R-CHOP Protocol

INTERVENTIONS:
Drug: Toripalimab, Rituximab — Toripalimab in combination with Rituximab will be administered every 3 weeks up to 4 cycles.
  Other Names: JS001, Rituximab
Drug: R-CHOP Protocol — After toripalimab plus rituximab treatment, R-CHOP regimen will be administered every 3 weeks in combination with R-CHOP up to 6 cycles.
  Other Names: Rituximab,Cyclophosphamide,Doxorubicin,Vincristine,Prednisone

SUMMARY:
1. Phase I portion of this study will evaluate the efficacy and saftey of toripalimab plus rituximab in treating untreated elderly diffuse large B cell lymphoma patients.
2. The aim of phase II portion of this study will evaluate the efficacy and saftey of toripalimab plus rituximab followed by R-CHOP(rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) regimen in treating untreated elderly diffuse large B cell lymphoma patients.

DETAILED DESCRIPTION:
The study consisted of a phase I and II portion. In phase I, patients accepted at least 2 cycles of toripalimab plus rituximab. Another 2 cycles of toripalimab plus rituximab will offered if they achieved CR. In phase II, all patients accpet R-CHOP regimen. If patient get CR after, they will accept 4 cycles of R-CHOP regimen, patients with PR,SD or PD will accept 6 cycles of R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
2. Aged 60-75 years old male or female;
3. Untreated,without any anti-lymphoma treatment;
4. DLBCL, or follicular lymphoma grade 3B, or transformed DLBCL, EBV (+) DLBCL, ALK (+) DLBCL, high-grade lymphoma were confirmed by histopathology examination;
5. Clinical stage II-IV, or stage I with bulky diesase (diameter > 7.5 cm);
6. International Prognostic Score (IPI): 2-5;
7. Paraffin tissue specimens or fresh puncture tissue specimens are available;
8. Eastern cooperative oncology group score: 0-2;
9. Estimated survival ≥ 12 months;
10. There must be at least one evaluate able or measurable lesion that meets the Lugano 2014 Lymphoma criteria [evaluable lesion: 18F-fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) examination showing increased lymph node or extranodal uptake (higher than liver) and PET and/or computed tomography (Computed Tomography) CT) features are consistent with lymphoma findings; lesions can be measured: nodular lesions > 15mm or extranodal lesions > 10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progress after radiotherapy), and accompanied by increased 18FDG uptake). Except for this, there is no measurable increase in diffuse 18FDG uptake in the liver;
11. Adequate organ and bone marrow function, no severe hematopoietic dysfunction, cardiac, pulmonary, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days prior to the use of the research drug): 1) The absolute value of neutrophils (>1.5×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 9 g/dL); 4) Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);
12. There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
13. Participants must pass a pulmonary function test (PFT) to confirm that forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is more than 60%, unless it is a large mediastinal mass caused by lymphoma that cannot meet this standard; carbon monoxide diffusion (DLCO), FEV1 and FVC are all above 50% of the predicted value; all PFT results must be obtained within four weeks before the first administration;
14. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within seven days before the first medication and the results are negative. WOBCP or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF until six months after the last dose of the research drug is used.

Exclusion Criteria:

1. Primary central nervous system lymphoma or secondary central nervous system involvement;
2. Hemophagocytic syndrome;
3. Previously treated with immunological checkpoint inhibitors (PD-1, PD-L1, CTLA-4, etc.);
4. History of severe allergies or allergic reactions to humanized or murine monoclonal antibodies;
5. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled;
6. Begin the study on subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a given condition within 14 days before treatment [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose) Sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens), except for tumor reduction due to large tumor burden (prednisone 30mg, bid × 5 days or equivalent dose of other glucocorticoid therapy);
7. In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix;
8. Begin the study and receive systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc.;
9. The study began with major surgery within 28 days before treatment or radiotherapy within 90 days before treatment;
10. Start the study and receive Chinese herbal medicine or Chinese patent medicine treatment within 7 days before treatment;
11. Begin research on live vaccination (except influenza attenuated vaccine) within 28 days before treatment;
12. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
13. Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group; 19. Patients with active pulmonary tuberculosis;
14. Start studying any active infections requiring systemic anti-infective treatment within 14 days of treatment.
15. Pregnant or lactating women;
16. People with known history of alcoholism or drug abuse;
17. Have uncontrollable complications, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or hemorrhagic diseases;
18. History of interstitial lung disease or non-infectious pneumonia. Subjects who had previously had non-infectious pneumonia caused by drugs or radiation but had no symptoms were allowed to enter the group;
19. The QTcF interval is more than 450 msec, unless it is secondary to bundle branch block;
20. Past psychiatric history; incapacitated or restricted;
21. According to the researchers' judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions;
22. Other researchers consider it unsuitable for patients to participate in this study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of toripalimab combined with Rituximab , Investigator-Assessed | upto 36 months
  Overall response was determined on the basis of investigator assessments according to the Lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET. Overall response was defined as the disappearance of all evidence of disease, regression of measurable disease, and no new sites.
The optimal dosage of Toripalimab combined with Rituximab | upto 6 months
  Maximum tolerable dose（MTD）and dose-limiting toxicity（DLT）of Toripalimab will be conducted in Phase Ib clinical studies. MTD and DLT is defined as protocol-defined Toripalimab related events.
Overall Response Rate (ORR) of toripalimab combined with Rituximab followed by R-CHOP regimen, Investigator-Assessed | upto 36 months
  Overall response was determined on the basis of investigator assessments according to the Lymphoma response to immunomodulatory therapy criteria (LYRIC) for Malignant Lymphoma, 2016. Tumor assessments were performed with CT/MRI with or without PET. Overall response was defined as the disappearance of all evidence of disease, regression of measurable disease, and no new sites.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Time from diagnosis until relapse or progression, non-protocol re-treatment of lymphoma, or death as a result of any cause, assessed up to 36 months
  Statistical analysis will entail descriptive statistics, and survival analysis including Kaplan-Meier estimates, log-rank testing of univariate prognostic factors, Cox proportional hazards analysis, as well as T-testing and regression analysis for comparing continuous variables in correlative study data.
Overall survival(OS) | OS is defined as the time from the treatment date to the death from any cause up to 60 months
  Statistical analysis will entail descriptive statistics, and survival analysis including Kaplan-Meier estimates, log-rank testing of univariate prognostic factors, Cox proportional hazards analysis, as well as T-testing and regression analysis for comparing continuous variables in correlative study data.
Percentage of Participants With Adverse Events (AEs) | Up to 36 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hematology department, Nanfang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No